CLINICAL TRIAL: NCT01368146
Title: Human Repeat Insult Patch Test of Wound Dressings
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Covalon Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TP-015
Record Dates: First submitted 2011-06-06; First posted 2011-06-07 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Skin Sensitization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- IV Clear™ (Experimental)
  Interventions: Device: IV Clear™
- Tegaderm CHG™ (Active Comparator)
  Interventions: Device: Tegaderm CHG™
- Control Vehicle Dressing (Placebo Comparator)
  Interventions: Device: Silicone Vehicle Control Dressing

INTERVENTIONS:
Device: IV Clear™ — Polyurethane film with a silicone adhesive dressing containing chlorhexidine and silver
  Arms: IV Clear™
Device: Tegaderm CHG™ — Polyurethane film with a polyacrylate adhesive and a polyol hydrogel containing 2% w/w chlorhexidine gluconate
  Arms: Tegaderm CHG™
Device: Silicone Vehicle Control Dressing — Polyurethane film with silicone adhesive dressing, without antimicrobials
  Arms: Control Vehicle Dressing

SUMMARY:
The purpose of this study is to determine whether contact sensitization occurs to the skin of normal healthy human subjects, by repetitive application of IV Clear™, Tegaderm CHG™ and Silicone Vehicle Control dressings.

DETAILED DESCRIPTION:
A single center, within-subject randomized study design in healthy adult subjects. Qualified subjects will complete three phases of the study (induction, rest and challenge).

Data for irritation, adhesion and pain upon removal will be collected from the individual patch sites.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years or older
* In good health, as determined by medical history and concomitant medication
* Able to comprehend and sign informed consent
* Unable to bear children or willing to use adequate birth control
* Willing and able to follow study directions, to participate in the study and to return for all specific visit

Exclusion Criteria:

* Subject pregnant, planning a pregnancy or lactating
* Diabetes (any type)
* Mastectomy involving removal of lymph nodes
* Clinically significant skin disease, including but not limited to psoriasis, eczema, atopic dermatitis, and active cancer
* Asthma or other severe respiratory disease requiring medication
* Self-reported immunological disorders including (but not limited to) HIV positive, AIDS, rheumatoid arthritis, and systematic lupus erythematosus
* Treatment of any type of cancer within the last two years or history of skin cancer in the test area
* Use of any of the following: topically applied products (e.g. medicals, lotions, creams, etc.) at the application site within 3 days of first application of test articles, immunosuppressive drugs within 30 days of first application of test articles, systemic or topical corticosteroids within 30 days of first application of test articles, and systemic or topically applied anti-inflammatory and antihistamine medications within 3 days of first application of test articles
* Participation in any patch test for irritation or sensitization within the last four weeks
* Participation in any investigational drug study within the last four weeks
* Damaged skin in or around the test sites which includes: sunburn, extremely deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or other disfiguration
* Known sensitization to adhesives, bandages, or materials used in test articles
* Medical condition which, in investigator's judgment, makes the subject ineligible or places the subject at undue risk

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Irritation | Assessed at induction phase (evaluated before reapplication; 9 applications over 3 weeks, reapplied after every 48 or 72 hrs) and challenge phase (single 48-hr application of test article to naive sites and evaluation 30 mins, 24 and 48 hrs post-removal
  Irritation assessed at the induction phase will be scored on a Berger and Bowman Scale. Irritation assessed at the challenge phase will be scored on a defined scale measuring erythema reactions, ranging from no reaction to strong erythema.

SECONDARY OUTCOMES:
Adhesion | Assessed at each 72 hour evaluation over three weeks, and once for a single 48-hour challenge application
  Adhesion was scored as follows:
  0 = no lift from skin (≥90% adherence)
  1. = some edges only lifting from skin (≥75% to ˂90% adherence)
  2. = less than half of the test article lifing (≥50% to ˂75% adherence)
  3. = more than half of the test article lifing but not detached (≥25% to ˂50% adherence)
  4. = test article detached (0% adherence)
Pain upon removal | Assessed by subjects at 72 hour evaluations over three weeks and a single 48-hour challenge application
  Any pain experienced during removal will be rated on a scale from 0 to 10, where 0 = no pain and 10 = worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Micah Humphrey, B.S., Principal Investigator — Hill Top Research
Locations (1):
- Hill Top Research, St. Petersburg, Florida, United States